CLINICAL TRIAL: NCT06825364
Title: Neural Responses to Tactile Auricular Stimulation Measured by Functional Near-infrared Spectroscopy in Pain-free Volunteers
Brief Title: Near-InfraRed Spectroscopy of Auricular Stimulation
Acronym: NIRAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Keith M Vogt, Associate Professor of Anesthesiology & Perioperative Medicine and Bioengineering, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY24090032
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Healthy Male and Female Subjects; Healthy Volunteer Study
Keywords: auricular stimulation; functional near infrared spectroscopy

STUDY DESIGN:
Intervention Model Description: Observational mechanistic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Auricular stim with fNIRS (Experimental): Points on the ear that correspond to the the shoulder, thumb, and lumbar spine (within an accepted cartography for auriculotherapy) will be stimulated repeatedly with flexible plastic (von Frey) filaments. A functional near-infrared spectroscopy cap will be worn, and brain responses to the stimulation will be recorded.
  Interventions: Other: auricular stimulation

INTERVENTIONS:
Other: auricular stimulation — Different points on both ears will be repeatedly stimulated with a plastic filament. This will be felt, but not be painful and should not result in lasting irritation.
  Other Names: von Frey filament

SUMMARY:
This is a single-visit non-invasive study of healthy volunteer subjects. Brain activity will be measured with infra-red light sensors attached to a cap worn on the head, while both ears are gently stimulated with plastic filaments.

DETAILED DESCRIPTION:
The aim of this study is to localize and quantify brain activations from experimental stimulation of auricular points in pain-free volunteers. Investigators will stimulate auricular points for the shoulder, thumb, and lumbar spine with von Frey filaments and measure functional near-infrared spectroscopy (fNIRS) responses in the primary somatosensory (S1) and prefrontal cortex (PFC). This will test the hypothesis that stimulation across different points in the auricular cartography maps to distinct brain responses, an assumption underpinning AT theory. Stimulation of different ear points is anticipated to induce similar PFC responses, but activate distinct areas within the S1 homunculus, validating the concept of auricular cartography.

ELIGIBILITY:
Inclusion Criteria:

Age of at least 18 years

Exclusion Criteria:

1. frequent or chronic pain requiring the use of pain-relieving medications more than twice per week, on average, in the last 3 months,
2. history or symptoms of neuropathy,
3. active lesions or skin disruptions to either ear,
4. recent (< 3 mo) illicit drug use,
5. history of substance misuse/abuse,
6. current or recent (<1 month) opioid or marijuana use, and
7. current regular use of psychoactive prescription medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
fNIRS response, Lumbar spine vs. thumb auricular points | 10 minutes
  Calculated T-statistic for contrast of analyzed fNIRS signal change, comparing responses from stimulation of the ipsilateral ear at the auricular points corresponding to the lumbar-spine vs. thumb.
  A T-statistic of 0 indicates no difference; more positive scores mean stronger fNIRS signal change with stimulation of the lumbar point, compared to stimulation of the thumb point; more negative scores mean change with stimulation of the thumb, compared to the lumbar spine. This outcome is a number reflecting the overall magnitude of difference between stimulation points, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.

SECONDARY OUTCOMES:
fNIRS response, shoulder vs. thumb auricular points | 10 minutes
  Calculated T-statistic for contrast of analyzed fNIRS signal change, comparing responses from stimulation of the ipsilateral ear at the auricular points corresponding to the shoulder vs. thumb.
  A T-statistic of 0 indicates no difference; more positive scores mean stronger fNIRS signal change with stimulation of the shoulder, compared to stimulation of the thumb point; more negative scores mean change with stimulation of the thumb, compared to the shoulder. This outcome is a number reflecting the overall magnitude of difference between stimulation points, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.
fNIRS response, lumbar spine vs. shoulder auricular points | 10 minutes
  Calculated T-statistic for contrast of analyzed fNIRS signal change, comparing responses from stimulation of the ipsilateral ear at the auricular points corresponding to the lumbar-spine vs. shoulder.
  A T-statistic of 0 indicates no difference; more positive scores mean stronger fNIRS signal change with stimulation of the lumbar point, compared to stimulation of the shoulder point; more negative scores mean change with stimulation of the shoulder, compared to the lumbar spine. This outcome is a number reflecting the overall magnitude of difference between stimulation points, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be publicly shared, after deidentification.
Time Frame: Individual participant data are anticipated to be available via open-access database within one year of study completion.